CLINICAL TRIAL: NCT04314596
Title: The Effects of Antioxidant Supplementation on Multiple Endurance Race Performance, Physiology, and Recovery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science & Performance Institute (Industry)
Collaborators: Lonza Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1219
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Oxidative Stress; Muscle Strength; Resistance Training; Body Composition; Muscle Damage
Keywords: Oxidative Stress; Muscle Strength; Resistance Training; Antioxidants

STUDY DESIGN:
Intervention Model Description: Double-Blind, parallel, randomized, placebo-controlled trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): Participants will engage in a one day, whole-body, cross-training course while consuming a visually identical placebo (25mg hydroxypropyl methylcellulose) 30 minutes prior to exercise on training days or with the first meal of the day on non-training days. Participants will then come in 24 and 48 hours post, cross-training course to be tested.
  Interventions: Other: Cross Training Course
- Experimental Group (Experimental): Participants will engage in a one day, whole-body, cross-training course while consuming the treatment condition (Oceanix™) 30 minutes prior to exercise on training days or with the first meal of the day on non-training days. Participants will then come in 24 and 48 hours post, cross-training course to be tested.
  Interventions: Other: Cross Training Course; Dietary Supplement: Oceanix

INTERVENTIONS:
Other: Cross Training Course — One day of a supervised, whole body, cross-training course that is meant to produce muscle damage and soreness.
Dietary Supplement: Oceanix — Ingredient contains highly active antioxidant enzymes, including superoxide dismutase (SOD), as well as essential fatty acids, vitamins, amino acids and minerals.
  Arms: Experimental Group

SUMMARY:
Thirty active male and female athletes will be recruited for the study. Subjects will be examined at baseline for VO2max performance. Subjects will then be stratified and randomly divided equally (50% - 50%) into an Oceanix (supplemental) or placebo condition such that baseline VO2max match. Once randomization, subjects will be baseline tested for multiple measures of muscle force capacity, muscle soreness, immune function, and endocrine function. Upon completion of baseline testing, subjects will all complete a one-day, cross-training course in Tampa, Florida. The training course is known to be extremely vigorous and causes significant muscle damage. Subjects will then be retested for muscle function at 24, and 48 hours following the course. At 24- and 48-hours subjects will be asked to repeat a simulated time trial race. In this way, we will measure repeated race performance, recovery from intense exercise, muscle damage from exercise, and immune function during multiple races.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18 to 45 years old
* At least one year of cross training experience (i.e. 3 days/week)

Exclusion Criteria:

* BMI of 30 or more kg/m²
* Any allergies to fish, shellfish, algae, or seaweed are excluded from participation
* Have any cardiovascular, metabolic, or endocrine disease
* Undergone surgery that affects digestion and absorption
* Smoking
* Drink heavily (> 7 and > 14 drinks per week for women and men, respectively)
* Women who are pregnant or planning to be pregnant
* Taking medication to control blood pressure, lipids, and blood glucose
* Have taken or currently taking anabolic-androgenic steroids

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Changes in muscle strength | Baseline, 24-Hour Post Cross-Training Course, 48-Hours Post Cross-Training Course.
  Assessed by isometric mid-thigh pull.
Changes in muscle power | Baseline, 24-Hour Post Cross-Training Course, 48-Hours Post Cross-Training Course.
  Assessed through ground reaction forces during countermovement and squat jumps on a force plate.
Changes in One(1) Mile Timed Run | Baseline, 24-Hour Post Cross-Training Course, 48-Hours Post Cross-Training Course.
  Experimental outcome assessing how quickly a 1 mile run can be completed.
Changes in Perceived Recovery Status (PRS) | Baseline, 1 Day of Cross-Training Course, 24-Hour Post Cross-Training Course, 48-Hours Post Cross-Training Course.
  Assessed through a visual analog scale (modified Borg Scale) numbered 0 to 10 with visual descriptors.
Changes in Rating of Perceived Exertion (RPE) | Baseline, 1 Day of Cross-Training Course, 24-Hour Post Cross-Training Course, 48-Hours Post Cross-Training Course.
  Assessed through a visual analog scale numbered 0 to 10 with visual descriptors.
Changes in Perceived Soreness Scale | Baseline, 1 Day of Cross-Training Course, 24-Hour Post Cross-Training Course, 48-Hours Post Cross-Training Course.
  Assessed through a visual analog scale numbered 0 to 10 with visual descriptors.

SECONDARY OUTCOMES:
Creatine Kinase | Baseline, 24-Hour Post Cross-Training Course, 48-Hours Post Cross-Training Course.
  Experimental outcome examining creatine kinase in fasted whole blood samples. This is biomarker an indirect measure of muscle damage.
Cortisol | Baseline, 24-Hour Post Cross-Training Course, 48-Hours Post Cross-Training Course.
  Experimental outcome examining the concentration of cortisol in fasted saliva samples.

OTHER OUTCOMES:
VO2max | Baseline
  Assessment of VO2max to determine fitness level and use as basis for randomization.

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Science & Performance Institute, Tampa, Florida, United States